CLINICAL TRIAL: NCT03184090
Title: An International, Non-controlled Phase II Trial to Identify the Molecular Mechanisms of Resistance and Sensitivity to Palbociclib Re-challenge Upon Progression to a Palbociclib Combination in ER-positive Metastatic Breast Cancer Patients
Brief Title: Molecular Mechanisms of Resistance and Sensitivity to Palbociclib Re-challenge in ER+ mBC
Acronym: BioPER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP089; 2015-003892-31 (EudraCT Number)
Record Dates: First submitted 2017-06-06; First posted 2017-06-12 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Palbociclib + Endocrine Therapy (Experimental): Patients will receive palbociclib capsules orally for 21 days every four weeks in combination with endocrine therapy (physician's choice based on prior administered agent including tamoxifen, exemestane, fulvestrant, anastrozole, or letrozole).
  Treatment will continue until disease progression (with the exception of patients who develop isolated progression in the brain), unacceptable toxicity, death, or discontinuation from the study treatment for any other reason.
  Interventions: Drug: Palbociclib; Drug: Endocrine therapy (non IMP)

INTERVENTIONS:
Drug: Palbociclib — palbociclib in combination with endocrine therapy (investigator's choice)
Drug: Endocrine therapy (non IMP) — Endocrine therapy (physician's choice based on prior administered agent including tamoxifen, exemestane, fulvestrant, anastrozole, or letrozole). Endocrine therapy must be different from previous treatment line.

SUMMARY:
This is an international, open-label, non-controlled, multicenter phase II clinical trial with two different primary objectives: a biological and a clinical objective.

From a clinical point of view, the objective is to assess the clinical benefit of the combination of palbociclib and hormonotherapy in patients with advance breast cancer that had previously received endocrine therapy in combination with palbociclib and had achieved clinical benefit during palbociclib treatment with subsequent disease progression.

From a biological point of view, the challenge is to define a molecular profile that allow identifying patients that could benefit more from continuing on palbociclib after progression on a prior palbociclib-containing regimen

DETAILED DESCRIPTION:
Eligible patients will receive palbociclib capsules orally for 21 days every four weeks in combination with endocrine therapy (physician's choice based on prior administered agent including tamoxifen, exemestane, fulvestrant, anastrozole, or letrozole).

Patients will receive treatment until disease progression (with the exception of patients who develop isolated progression in the brain), unacceptable toxicity, death, or discontinuation from the study treatment for any other reason.

Patients discontinuing the study treatment period will enter a post-treatment follow-up period during which survival and new anti-cancer therapy information will be collected every six months (± 14 days) from the last dose of investigational product. The treatment follow-up period will conclude at six months after the last patient has received first treatment dose in the study.

ELIGIBILITY:
Inclusion Criteria:

* Pre- and postmenopausal women age ≥ 18 years (Premenopausal women must be treated with LHRH analogues for at least 28 days prior to study entry)
* Hormone receptor-positive [estrogen receptor (ER) and/or progesterone receptor (PR)] and HER2-negative
* Locally advanced or mBC that had previously received no more than two prior lines of endocrine therapy and no more than one prior line of chemotherapy for advanced disease.
* Inmmediate previous treatment with palbociclib in combination with endocrine therapy had achieved clinical benefit during palbociclib-based treatment
* Evidence of measurable and biopsable metastatic disease is required
* Confirmed disease progression on immediate previous palbociclib plus endocrine therapy.
* Last dose of palbociclib administered no later than eight weeks and not earlier than three weeks from study entry.
* No prior use of at least one of the reasonable endocrine therapy options: tamoxifen, fulvestrant, letrozole/anastrozole, or exemestane.
* Patients agree to collection of blood samples (liquid biopsy) and collection of metastatic tumour sample (biopsy) at the time of inclusion and progression (if appropriate).
* Adequate organ function.
* Resolution of all acute toxic effects of prior anti-cancer therapy or surgical procedures

Exclusion criteria

* HR or HER2 unknown disease.
* HER2-positive disease based on local laboratory results [performed by immunohistochemistry/fluorescence in situ hybridization (FISH)].
* Locally advanced breast cancer candidate for a local treatment with a radical intention.
* Formal contraindication to endocrine therapy.
* Progressing central nervous system (CNS) disease.
* Patients with exclusive non-measurable/evaluable disease.
* Other malignancies within the past five years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix.
* Major surgery (defined as requiring general anaesthesia) or significant traumatic injury within four weeks of start of study drug, or patients who have not recovered from the side effects of any major surgery, or patients that may require major surgery during the course of the study.
* Patients with an active bleeding diathesis, previous history of bleeding diathesis, or anti-coagulation treatment (the use of low molecular weight heparin is allowed as soon as it is used as prophylaxis intention).
* Have a serious concomitant systemic disorder (i.e., active infection including HIV, or cardiac disease) incompatible with the study (at the discretion of investigator).
* Are unable to swallow tablets.
* History of malabsorption syndrome or other condition that would interfere with enteral absorption.
* Chronic daily treatment with corticosteroids with a dose of ≥10 mg/day methylprednisolone equivalent (excluding inhaled steroids).
* QTc >480 msec on basal assessments, personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation, or Torsade de Pointes (TdP).
* Uncontrolled electrolyte disorders that can compound the effects of a QTc-prolonging drug (i.e., hypocalcemia, hypokalemia, or hypomagnesemia).
* Known hypersensitivity to any palbociclib excipients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2020-10-27 (Actual)

PRIMARY OUTCOMES:
molecular patterns of resistance [with a special focus on retinoblastoma (Rb) status] upon progression to palbociclib plus endocrine therapy in patients who previously achieved clinical benefit with the combination | Baseline-Up to 24 months
  the percentage of patients with Rb loss [as defined by loss of expression, copy number variation (CNV), somatic mutation, or methylation dependent silencing]. The evaluation criteria will be the characterization of the molecular patterns of resistance with greater than 20% prevalence.
clinical activity of the combination of palbociclib and endocrine therapy after prior progression to palbociclib in endocrine-sensitive patients. | Baseline-Up to 24 months
  percentage of patients that achieve clinical benefit (CBR) defined as complete response, partial response, or stable disease for at least 24 weeks per RECIST v.1.1.

SECONDARY OUTCOMES:
Compare clinical activity with molecular patterns of resistance. | Baseline-Up to 24 months
  Patients with molecular patterns of resistance (Rb loss, biomarkers significant inhibition), mutations and expression profiles will be compared against patients without.
Measure changes of immunostaining of Rb targets (E2F, DNMT, HIF1alpha, and SKP2) as a result of CDK4 and CDK6 inhibition and the potential predictive value of cyclin D, cyclin E, p16, p18, p21, and p27, in CDK4, and CDK6 inhibition | Baseline-Up to 24 months
  measure histoscore (Hscore) levels of the above targets

OTHER OUTCOMES:
Measure senescence and apoptosis (Ki67 and active caspase 3) in subgroups of patients with varying clinical responses. | Baseline-Up to 24 months
  Measure histoscore (Hscore) levels of Ki67 and active caspase 3
Measure differences in expression profile, assessed by RNA microarrays | Baseline-Up to 24 months
  Differences in expression profiles, assessed by RNA microarrays.
Correlation between inhibitory effects of palbociclib and clinical response | Baseline-Up to 24 months
Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs grade 3 and 4 and Serious Adverse Events) | Baseline-Up to 24 months
Compare inhibitory effects of palbociclib and clinical response in patients with visceral disease or patients who received prior (neo) adjuvant hormonal therapy | Baseline-Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Javier Cortes, MD PhD, Principal Investigator — Hospital Universitario Ramon y Cajal
Locations (15):
- Italy (2):
  - Istituto Europeo di Oncologia, Milan
  - Azienda Sanitaria Universitaria Integrata di Udine, Udine
- Spain (13):
  - ICO Badalona, Badalona, Barcelona
  - ICO l'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Clinico Universitario A Coruña, A Coruña
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Provincial de Castellón, Castellon
  - Hospital Reina Sofia, Córdoba
  - Hospital La Paz, Madrid
  - Hospital Sant Joan de Reus, Reus
  - Hospital Virgen del Rocío, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Instituto Valenciano de Oncología - IVO, Valencia

IPD SHARING:
Plan to Share IPD: No